CLINICAL TRIAL: NCT04606394
Title: Peak Inspiratory Flow (PIF) and Dry Powder Inhaler (DPI) Performance in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Peak Inspiratory Flow and Dry Powder Inhaler Performance in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pulmonary Research Institute of Southeast Michigan (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2020-10-19; First posted 2020-10-28 (Actual); Results first posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2020-12

CONDITIONS: COPD
Keywords: DPI; PIF; FEV1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: Open label comparative design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open label treatment (Other): All subjects receive Trelegy and Ventolin for 2 weeks
  Interventions: Drug: Trelegy Ellipta 100/62.5/25Mcg Inh 30D; Drug: Ventolin 90Mcg/Actuation Inhalation Aerosol

INTERVENTIONS:
Drug: Trelegy Ellipta 100/62.5/25Mcg Inh 30D — Administration of Trelegy in all patients
  Other Names: DPI Delivery
Drug: Ventolin 90Mcg/Actuation Inhalation Aerosol — 2 hours after the administration of Trelegy, administer Ventolin in all patients
  Other Names: pMDI Delivery

SUMMARY:
The purpose of the study is to determine whether PIF is clinically important when using the Ellipta DPI device. In addition, the study will validate the best/most clinically appropriate way to perform a PIF maneuver, to determine the testing capabilities of the preferred PIF maneuver and to relate this PIF measurement to meaningful clinical outcomes in COPD patients

DETAILED DESCRIPTION:
Study Design and Methods Rationale

* The expected FEV1 response to a bronchodilator is uncertain as multiple factors influence this measure, including severity of disease, day to day variability, varying reversibility in COPD patients, the delivery of the drug to a patient and the effectiveness of the medication delivered. Thus, the measurement of an acute bronchodilator response after delivering a long acting bronchodilator may not identify whether a medication has been effectively delivered to a patient.
* However, if a long acting bronchodilator has not been effectively delivered to the lung, then subsequent delivery of a short acting bronchodilator should produce a significant additional bronchodilator response. On the other hand, if a long acting bronchodilator has been effectively delivered to the lung, then subsequent delivery of a short acting bronchodilator should not produce any further significant bronchodilation.
* Based on this rationale, comparison of the acute bronchodilator response to a short acting bronchodilator after receiving a long acting should identify whether drug delivery is ineffective in a selected patient population, irrespective of baseline FEV1 and of any partial response to the long acting bronchodilator. Comparison of the short acting bronchodilator measurement between patient groups with differing PIF thresholds should identify whether PIF has an impact of drug delivery of a long acting bronchodilator via a DPI.
* Open label design comparing the acute bronchodilator response after delivery of a long acting bronchodilator via Ellipta DPI in patients with normal, suboptimal and minimal PIF.

ELIGIBILITY:
Inclusion Criteria:

* smoking history >10 pack years
* pre-bronchodilator FEV1 <60% predicted
* post-bronchodilator FEV1/FVC <70%
* female participants are eligible to participate if they are not pregnant, not breastfeeding, and at least one of the following conditions applies:
* not a woman of childbearing potential OR
* agree to follow the contraceptive guidance during the treatment period and until the safety follow-up contact after the last dose of study treatment
* stratification requiring at least 1/3 of patients having a PIF of < 60L/min (AM pre-dose based on using the level 2 InCheck Dial resistance setting with a sharp maximal effort starting after exhaling fully)

Exclusion Criteria:

* any subject with unstable disease, including
* COPD exacerbation in the last 6 weeks
* upper respiratory tract in in the last 4 weeks
* COPD or upper respiratory tract infection during run-in (subjects may be re-screened x 1 when stable after an acute event)
* pulmonary disease other than COPD
* any lung resection
* unstable cardiac conditions (at the discretion of the investigator)
* other unstable medical conditions (at the discretion of the investigator)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary T Ferguson, MD, Principal Investigator — Pulmonary Research Institute of Southeast Michigan
Locations (1):
- Pulmonary Research Institute of Southeast Michigan, Farmington Hills, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perugini V, Rhee CK, Moon JY, Pei Yee T, Ra SW, Pirina P, Yoo KH, Navarrete BA, Gouder C, Pacheco A, Navarro-Rolon A, Harlander M, Lapperre T, Loh SCH, Fole D, Naval E, Palacios PJR, Miravitlles M, Usmani O. Assessment of peak inspiratory flow in patients with chronic obstructive pulmonary disease: a multicentre, observational, prospective, real-life study. BMJ Open Respir Res. 2025 Sep 25;12(1):e002408. doi: 10.1136/bmjresp-2024-002408. PMID 40998461

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Severe/very severe COPD patients in stable condition stratified to insure that at least 12 of 30 subjects had a suboptimal peak inspiratory flow (PIF <60L/min)
Pre-assignment Details: Enrollment, run-in on current maintenance therapy followed by testing, conversion of maintenance therapy to Trelegy Ellipta therapy for 2 weeks followed by testing
Groups:
- Trelegy Ellipta Open Label Treatment: All subjects receive Trelegy and Ventolin for 2 weeks
  Trelegy Ellipta 100/62.5/25Mcg Inh 30D: Administration of Trelegy in all patients
  Ventolin 90Mcg/Actuation Inhalation Aerosol: 2 hours after the administration of Trelegy, administer Ventolin in all patients
Period: Overall Study
Arm/Group | Trelegy Ellipta Open Label Treatment
Started | 45 (45 subjects recruited/consented. 12 failed entry criteria during screening and 3 withdrew consent during screening for non-medical reasons. 30 subjects met entry criteria per protocol and started/completed the study.)
Completed | 30
Not Completed | 15
Not completed — Withdrawal by Subject | 3
Not completed — Exclusion criteria screen failure | 12

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Using triple therapy at baseline [Count of Participants; unit: Participants] | 18
CAT score ≥10 [Count of Participants; unit: Participants] — COPD Assessment TesT (CAT) - Quality of Life Health Assessment Tool - range from 0-40, with a higher number identifying more severe symptoms. CAT score of 10 or higher used to define a symptomatic COPD patient.
  Participants | 30
CAT score ≥15 [Count of Participants; unit: Participants] — COPD Assessment TesT (CAT) - Quality of Life Health Assessment Tool - range from 0-40, with a higher number identifying more severe symptoms. CAT score of 15 or higher used to define a very symptomatic COPD patient.
  Participants | 28
History of 2 moderate/1 severe exacerbation [Count of Participants; unit: Participants] | 9
History of severe exacearbtion [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: DPI Responder Analysis in Patients With Suboptimal PIF (<60 L/Min)
Description: Outcome = the number of subject test days (2 test days per subject) meeting responder criteria defined as:
  DPI Responder - a positive (>50 ml) peak FEV1 response 2 hours after Trelegy Ellipta® DPI with a negative (<50mL) peak FEV1 response 30 minutes after Ventolin® pMDI (2.5 hours post Trelegy) DPI Partial Responder a positive (>50 ml) peak FEV1 response 2 hours after Trelegy® Ellipta DPI with a positive (>50 ml) peak FEV1 response 30 minutes after Ventolin® pMDI (2.5 hours post Trelegy) DPI Failure - a negative (<50mL) peak FEV1 response 2 hours after Trelegy Ellipta® DPI with a positive (>50 ml) peak FEV1 response 30 minutes after Ventolin® pMDI (2.5 hours post Trelegy) Irreversible - a negative (<50mL) peak FEV1 response 2 hours after Trelegy Ellipta® DPI with a negative (<50mL) peak FEV1 response 30 minutes after Ventolin® pMDI (2.5 hours post Trelegy)
Time Frame: 2 weeks
Population: Number of subject test days (2 per subject) with DPI Failure based on baseline PIF <60 L/min or >60 L/min
Measure: Number; unit: Number of subject test days
Units Other Than Participants: Subjet test days
Groups:
- Suboptimal PIF: Subject with PIF < 60 L/min at baseline
- Normal PIF: Subjects with PIF > 60 L/min at baseline
Arm/Group | Suboptimal PIF | Normal PIF
Number analyzed (Participants) | 12 | 18
Number analyzed (Subjet test days) | 24 | 36
Number of subject test days | 2 | 1
Statistical Analysis 1: Comparison: Suboptimal PIF vs Normal PIF; Data outcome reported was the number and percentage of subject test days with DPI Failure in subjects in suboptimal PIF (<60 L/min) versus normal PIF subjects. Statistical analysis performed was a comparison between rates of DPI Failure in the 2 groups; Test type: Superiority; p = 0.33, Chi-squared; Mean Difference (Final Values) = 1

2. Secondary Outcome: DPI Responder Analysis in Patients With Reduced PIF (<45 L/Min)
Description: as for outcome 1
Time Frame: 2 weeks
Population: Number of subject test days (2 per subject) with DPI Failure based on baseline PIF <45 L/min or >45 L/min
Measure: Number; unit: Number of subject test days
Units Other Than Participants: Number of sub ject test days
Groups:
- Reduced PIF: PIF <45 L/min at baseline
- Normal PIF: PIF > 45 L/min at baseline
Arm/Group | Reduced PIF | Normal PIF
Number analyzed (Participants) | 6 | 24
Number analyzed (Number of sub ject test days) | 12 | 48
Number of subject test days | 2 | 1
Statistical Analysis 1: Comparison: Reduced PIF vs Normal PIF; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.04, Chi-squared; Mean Difference (Final Values) = 1

3. Secondary Outcome: PIF Measurement Techniques
Description: PIF value (L/min) based on different PIF measurement techniques
Time Frame: Baseline on day of testing
Population: All subjects
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Ellipta PIF Standing: Performance of PIF using Ellipta instructions while standing
- Ellipta PIF Sitting: Performance of PIF using Ellipta instructions while sitting
- Instructed PIF: Pif measured with maximal PIF instrucitons only
- Encouraged PIF: Pif measured while instructed and encouraged for maximal effort
- Spiro PIF: PIF measured with maximal inspiratory effort/flow loop during spirometry
Arm/Group | Ellipta PIF Standing | Ellipta PIF Sitting | Instructed PIF | Encouraged PIF | Spiro PIF
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30
L/min | 52 (17) | 53 (25) | 70 (18) | 74 (18) | 137 (67)

ADVERSE EVENTS:
Time Frame: 6 weeks - from consent to 1 week post completion of study
Description: No difference in definitions
Arm/Group | Open Label Treatment
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

LIMITATIONS AND CAVEATS:
No primary information was available to derive power calculations to estimate the number of subjects needed to test the study hypothesis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT04606394/Prot_SAP_ICF_001.pdf